CLINICAL TRIAL: NCT02968472
Title: Single Center, Open, Phase I Clinical Trial of 4SCAR19 Cells in the Treatment of Relapsed and Refractory B Cell Leukemia
Brief Title: A Phase I Trial of 4SCAR19 Cells in the Treatment of Relapsed and Refractory B Cell Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Yunnan (Other)
Collaborators: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Xun Lai, chief physician, The First People's Hospital of Yunnan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXUN
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: B Acute Lymphoblastic Leukemia
Keywords: 4s CAR-T19; B cell leukemia; B-ALL
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- prophylactic 4SCAR19 cells (Experimental): Patients who have relapsed and refractory B cell leukemia after chemotherapy will be treated prophylactically with CD19-specific gene-engineered T cells.
  Interventions: Genetic: prophylactic 4SCAR19 cells

INTERVENTIONS:
Genetic: prophylactic 4SCAR19 cells — Autologous 4th generation withdrawal lentiviral-transduced 4S CAR-T19

SUMMARY:
A chimeric antigen receptor gene-modified T cells (CART: 4SCAR19)by targeted the CD19 (cluster of differentiation antigen 19), treat patients with CD19 positive malignant B cells tumor, assess treatment safety, and observe therapeutic effects. At the same time,the change process of the CART and residual tumor status of the patient are observe dynamically， which summarizes the best therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 6 months.
* the immune phenotype analysis of patients with malignant B cell surface expression CD19 molecules.
* the Karnofsky performance status score over 80 points, is expected to patients survival time is more than 3 months.
* the important viscera function meet: heart ultrasound tip heart ejection fraction 50% or higher, electrocardiogram (ecg) not seen obvious abnormality;The blood oxygen saturation 90% or higher;Creatinine 2.5 times normal range or less; aspartate aminotransferase and aspartate aminotransferase3 times normal range or less, total bilirubin of 2.0 mg/dl or less.
* or greater Hgb 80 g/L.
* no contraindications to solid and cell separation
* the patient and family to have a strong willingness to participate in clinical trials, and are willing to bear all the consequence caused by the test failed, and sign the informed consent.
* the panel discussion, combined with patient general condition, think the benefit is greater than the risks involved in the clinical trials.

Exclusion Criteria:

* accompanied with other active disease, the treatment is difficult to correct.
* bacteria, fungus, or virus infection, unable to control.
* people living with HIV.
* active hepatitis B virus and hepatitis C virus infection.
* of pregnancy and nursing mothers.
* before entering the test of the use of glucocorticoid systemic treatment within a week.
* confirmed before used CAR - but invalid patients treated T cells, after in the physical examination, experts discuss confirmed by a team doesn't fit in the CAR again - T treatment.Before used gene therapy method.
* the researchers believe that might increase risk subjects or interfere with the test results of any situation.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Safety Using CTCAE 4 standard to evaluate the level of adverse events after receiving the cells. | 24 weeks
  Safety of fourth generation anti CD19 CAR-T cells in patients with relapsed and refractory B-ALL - Using CTCAE 4 standard to evaluate the level of adverse events after receiving the cells.

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation anti CD19 CAR-T cells in patients with relapsed or refractory B-ALL (B cell acute lymphoblastic leukemia) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Huang Jianzhang, Doctor, Study Chair — Shenzhen immune gene therapy research institute
Locations (1):
- First people's hospital of Yunnan province, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai X, Sun YY, Chang LJ, Ma YR, Gu XZ, Yao XM, Nie B, Wen Y, Zhang XM, Jiang YX, Yang H, Yu LQ, Fang MJ, Wang L, Yuan Bo X. Could cytokine release syndrome induce acute myelofibrosis in CD19 chimeric antigen receptor T cells therapy? Bioengineered. 2020 Dec;11(1):824-828. doi: 10.1080/21655979.2020.1791597. PMID 32772769